CLINICAL TRIAL: NCT00617227
Title: Measurement of Serum Vancomycin in Patients Receiving Enteral ( Oral/Intracolonic) Vancomycin.
Brief Title: Serum Vancomycin Levels in Patients Receiving Enteral Vancomycin
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Edward K.Chapnick, MD Director Division of Infectious Diseases, Maimonides Medical Center
Other Study IDs: Maimid; Resident research grant
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Clostridium Difficle Colitis; Clostridium Difficle Associated Disease
Keywords: Enteral vancomycin therapy, serum vancomycin levels, renal failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is based on the hypothesis that decreased creatinine clearance may be associated with detectable vancomycin levels in patients on enteral (oral / vancomycin enemas) vancomyicn for CDAD.

The objective of the study is to see whether enteral vancomycin is absorbed through the inflamed GI mucosa in CDAD, and if it is absorbed, does it achieve measurable serum concentration.

DETAILED DESCRIPTION:
Vancomycin is a large glycopeptide compound with a molecular weight of about 1450 Da. It is not appreciably absorbed orally and is eliminated primarily via the renal route. Enteral vancomycin therapy (oral/intracolonic ) is used inpatients with severe Clostridium difficile associated colitis who are unable to take oral metronidazole or have failed treatment with metronidazole. Oral vancomycin is not detectable in serum of normal persons, but concentrations below therapeutic range may be found in patients with colitis. There are a few case reports of serum concentrations within the therapeutic range after oral/intracolonic administration of vancomycin, in association with renal failure. The use of enteral vancomycin in our geriatric population with variable creatinine clearance prompted us to measure the serum vancomycin levels in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients on enteral vancomycin therapy

Exclusion Criteria:

* Coadministration of intravenous vancomycin therapy,intravenousvancomycin administration in previous10 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Clostridium difficile associated colitis on enteral vancomycin therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Patients with detectable serum vancomycin levels during enteral vancomycin therapy | 5-7days

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Chapnick, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States